CLINICAL TRIAL: NCT02871947
Title: Epidemiology and Cytokines Analysis of Severe Asthma Patients in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Diahn-Warng Perng, Department of Chest Medicine, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2016-03-010AC
Record Dates: First submitted 2016-08-16; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-03

CONDITIONS: Bronchial Asthma; Cytokines
Keywords: severe asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe asthma is a heterogeneous disease characterized by the need for treatment with high doses of inhaled corticosteroids. It affects 5%-10% of asthmatic patients, although it accounts for a significant percentage of the consumption of health care resources. Severe asthma comprises various clinical and pathophysiological phenotypes. In this current study, we aimed to clinical characteristics and cytokes profile in severe asthma patients.

DETAILED DESCRIPTION:
To investigate the clinical phenotypes and inflammatory endotype by analyzing cytokines in severe asthma patients, it may improve characterization of the disease and contribute to improved selection of appropriate treatment. It could also help link genotypes with their phenotypic manifestations and their natural history and prognosis. A greater understanding of the phenotypes of severe asthma could enable identification of biomarkers for each phenotype, and identify the association between biokarkers and clinical outcomes in severe asthma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Asthma which requires treatment with guidelines suggested medications for GINA steps 4-5 asthma (high dose ICS and LABA or leukotriene modifier/theophylline) for the previous year or systemic CS for 50% of the previous year to prevent it from becoming ''uncontrolled'' or which remains ''uncontrolled'' despite this therapy
2. Uncontrolled asthma defined as at least one of the following:

(1). Poor symptom control: ACQ consistently>1.5, ACT<20 (or ''not well controlled'' by NAEPP/GINA guidelines) (2). Frequent severe exacerbations: two or more bursts of systemic CS (>3 days each) in the previous year (3). Serious exacerbations: at least one hospitalization, ICU stay or mechanical ventilation in the previous year (4). Airflow limitation: after appropriate bronchodilator withhold FEV1<80% predicted (in the face of reduced FEV1/FVC defined as less than the lower limit of normal)

Exclusion Criteria:

* (1). mild to moderate persistent asthma (2). COPD or other lung diseases (3). malignancy (4). long-term O2 therapy more than 15 hours/day (5). long-term NIPPV use (> 6 hours/day) (6). no inform consent and cannot be followed regularly (7). active TB or other infection diseases

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: severe asthma patients who have received high-dose ICS and still being not well controlled
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
asthma acute exacerbation | 1 year follow-up

SECONDARY OUTCOMES:
inflammatory biomarkers | 1, 3, 6, 9. 12 months
  IgE and Eosphile count

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Veterans Genral Hospital, Taipei, Taiwan
  - Chest department, Veteran General Hospital-TAIPEI, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No